CLINICAL TRIAL: NCT07045714
Title: Bilateral Lumbar Decompression Via Uniportal Endoscopic Laminotomy in Patients With Lumbar Spinal Stenosis: Multicentric Case Series
Acronym: MELD-1
Status: Not yet recruiting | Type: Observational
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: Tecnologico de Monterrey (Other); Centro Medico Nacional Siglo XXI IMSS (Other); Hospital Ángeles Tijuana (Unknown); Hospital Zambrano Hellion TecSalud, Mexico (Unknown); TecSalud (Unknown)
Responsible Party: Sponsor
Other Study IDs: MELD-1
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Lumbar Spinal Stenosis; Minimally Invasive Surgical Procedures; Endoscopic Spine Surgery; Spinal Degenerative Disease
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar Spinal Stenosis Cases: Patients diagnosed with lumbar spinal stenosis who exhibit persistent neurological deficits and pain despite receiving at least three months of conservative treatment. All participants have elected to undergo ULBLD using endoscopic uniportal technique. They are being prospectively followed to evaluate improvements in neurological function and reductions in pain-related disability, as well as to document perioperative outcomes including surgical time, blood loss, hospital stay, and complications.
  Interventions: Procedure: Unilateral Laminotomy with Bilateral Lumbar Decompression (ULBLD)

INTERVENTIONS:
Procedure: Unilateral Laminotomy with Bilateral Lumbar Decompression (ULBLD) — Unilateral laminotomy with bilateral lumbar decompression (ULBLD) using endoscopic uniportal technique

SUMMARY:
Lumbar spinal stenosis is a condition that can cause pain, sensory disturbances, and motor deficits due to the compression of neural structures in the lumbar spine. While conservative treatments such as physical therapy and pain management can help some patients, others with persistent neurological deficits may require surgical intervention. Traditional surgical approaches, including open laminectomy, have proven effective but carry risks such as extensive muscle damage, considerable blood loss, postoperative spinal instability, and prolonged recovery times.

This study evaluates a minimally invasive surgical approach called unilateral laminotomy with bilateral lumbar decompression (ULBLD) using endoscopic uniportal technique as an alternative to traditional methods for patients with lumbar spinal stenosis. The main objective is to assess changes in neurological deficits and disability in patients with lumbar spinal stenosis following this procedure. The study will also document hospitalization duration, surgical time, blood loss, and the incidence of postoperative complications.

This multicenter, prospective case series will recruit 78 patients from three medical centers in Mexico. Participants must have symptomatic lumbar spinal stenosis that persists despite at least three months of conservative treatment. Eligible patients will undergo ULBLD using endoscopic uniportal technique, a method that allows precise nerve decompression through a small incision, minimizing damage to surrounding tissues. Standardized clinical assessment tools, including the Japanese Orthopaedic Association (JOA) scale for lumbar disease, Oswestry Disability Index (ODI), and Visual Analog Scale (VAS) for pain, will be used to evaluate outcomes at multiple time points over 12 months.

By comparing patients' preoperative and postoperative evaluations, the study aims to determine whether ULBLD using endoscopic uniportal technique effectively improves neurological function and reduces disability while maintaining a favorable safety profile. Findings from this study could lead to a more precise understanding of the impact of ULBLD on disability, pain, and health-related quality of life for patients with lumbar spinal stenosis.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a common degenerative condition characterized by narrowing of the lumbar spinal canal, resulting in compression of nerve roots and, in some cases, the spinal cord. This narrowing can be caused by degenerative changes such as hypertrophy of the ligamentum flavum, formation of osteophytes, intervertebral disc protrusion, and thickening of the facet joints. Although its prevalence increases with age, it can affect people of different age groups. Clinically, patients present symptoms such as lumbar pain, neurogenic claudication, paresthesias, and weakness in the lower extremities, which significantly decrease their quality of life. These symptoms limit the ability to perform daily activities and reduce functional independence, affecting the general well-being of individuals.

This study investigates the use of ULBLD using endoscopic uniportal technique, a minimally invasive surgical approach that offers targeted decompression through a single small incision while minimizing tissue disruption. The primary objective of the study is to evaluate changes in neurological deficits and disability in patients with lumbar spinal stenosis following this procedure. Secondary objectives include assessing the duration of hospitalization, surgical time, blood loss, and the incidence of postoperative complications.

This multicenter, prospective case series will recruit 78 patients diagnosed with lumbar spinal stenosis at three medical institutions in Mexico. The study will be conducted over a period of 24 months, with an initial 12-month patient recruitment phase, followed by postoperative follow-up assessments at predetermined time intervals up to one year. Participants will undergo ULBLD using endoscopic uniportal technique, a method designed to preserve spinal mobility while reducing compression on the nerve roots. The procedure will be performed under general anesthesia with continuous neurophysiological monitoring, including somatosensory evoked potentials, motor evoked potentials, and continuous electromyography. Using a working-channel endoscope, surgeons will perform laminotomies to remove compressive elements such as osteophytes, hypertrophic ligaments, or herniated disc material. The technique is aimed at achieving decompression with minimal disruption to the surrounding soft tissues.

Patients must meet specific inclusion criteria, including an age range of 18 to 75 years, confirmed diagnosis of lumbar spinal stenosis (Lee classification grade I-III), and the presence of neurological symptoms unresponsive to at least three months of conservative management. Exclusion criteria include prior lumbar surgery at the affected level, active infections, systemic inflammatory diseases, vertebral instability, congenital spinal malformations, and contraindications for general anesthesia.

Patient outcomes will be systematically evaluated using validated clinical assessment tools, including:

* Japanese Orthopaedic Association (JOA) Scale for lumbar disease to assess neurological function and functional status.
* Oswestry Disability Index (ODI) to measure the impact of lumbar pain on daily activities.
* Visual Analog Scale (VAS) for pain to quantify lumbar and lower limb pain intensity.
* EQ-5D-5L health-related quality of life questionnaire to evaluate overall well-being.
* Modified MacNab Criteria to determine patient satisfaction with surgical outcomes.

Descriptive statistical methods will be used to analyze demographic and clinical characteristics of the study population. Changes in primary and secondary outcomes will be evaluated using paired ttests for continuous variables and Chi-square tests for categorical variables. The impact of the procedure on neurological function and pain relief will be assessed through longitudinal comparisons between baseline and follow-up assessments at 1, 3, 6, and 12 months postoperatively. The incidence of complications will be categorized using the Clavien-Dindo classification, and the Comprehensive Complication Index will be used to quantify cumulative morbidity.

This study complies with the Declaration of Helsinki, the International Council for Harmonisation Good Clinical Practice (ICH-GCP) guidelines, and national regulatory requirements. All participants will provide written informed consent before enrollment, and patient confidentiality will be maintained through data pseudonymization. The study has been approved by the Ethics Committees of the participating institutions.

The expected impact of this study is to generate clinical evidence supporting ULBLD using endoscopic uniportal technique as a safe and effective alternative to traditional surgical approaches for lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent to participate in the study.
* Age ≥18 years and <75 years.
* Patients with lumbar spinal stenosis grade I-III according to the Lee scale.
* Radicular or myelopathic symptoms.
* Having undergone complete conservative management, including physical therapy and analgesia, for at least 3 months.
* Patients who have opted for ULBLD using endoscopic uniportal technique for lumbar spinal stenosis.

Exclusion Criteria:

* Inability to read or write.
* Prior lumbar surgeries at the levels to be treated.
* Infectious symptoms or concomitant rheumatologic diseases.
* Criteria of lumbar vertebral instability.
* Congenital spinal malformations.
* Disc herniation at the same lumbar level to be operated on.
* Medullary hyperintensity on T2-weighted magnetic resonance imaging in the levels to be treated.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar spinal stenosis who continue to experience symptoms despite receiving complete conservative management for at least 3 months and who have chosen to undergo ULBLD using endoscopic uniportal technique will be recruited consecutively. Recruitment will take place at the following healthcare centers:
  * Centro Médico Zambrano-Hellion, TecSalud (San Pedro Garza García, N.L.) and Clínica Cuauhtémoc y Famosa (Monterrey, N.L.). Patients will be recruited by Dr. Mario Benvenutti Regato, a neurosurgery specialist with over 7 years of experience performing endoscopic spine surgery.
  * Centro Médico Nacional Siglo XXI (Mexico City)Patients will be recruited by Dr. Félix Domínguez Cortinas, a neurosurgery specialist with over 10 years of experience performing endoscopic spine surgery.
  * Hospital Ángeles Tijuana (Tijuana, B.C.)Patients will be recruited by Dr. Alfonso García Chávez, a specialist in traumatology and orthopedics with over 10 years of experience
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Lumbar Disability (Oswestry Disability Index) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure assesses disability related to lumbar pain using the Oswestry Disability Index (ODI), a validated instrument scored from 0% (no disability) to 100% (maximum disability). It quantifies the impact of lumbar pain on daily activities and overall function. Changes in ODI scores over time will reflect the effectiveness of the surgical intervention in reducing pain-related disability.
Change in Neurological Function (Japanese Orthopaedic Association Score for Lumbar Disease) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure evaluates neurological function using the Japanese Orthopaedic Association (JOA) scale for lumbar disease. The JOA score, which ranges from -6 to 29 points (where higher scores indicate better neurological function), assesses lumbar pain, lower extremity pain and walking capacity, clinical signs, and restriction in activities of daily living. Improvements in the JOA score following surgery will be used as an indicator of enhanced neurological status.

SECONDARY OUTCOMES:
Change in Back Pain Intensity (Visual Analog Scale - Back) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure assesses the intensity of back pain using the Visual Analog Scale (VAS) for back pain, a validated instrument where patients mark their level of pain on a horizontal line from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst imaginable pain". Changes in VAS-back scores over time will reflect the effectiveness of the surgical intervention in reducing back pain intensity.
Change in Lower Extremity Pain Intensity (Visual Analog Scale - Lower Extremity) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure assesses the intensity of lower extremity pain using the Visual Analog Scale (VAS) for lower extremity pain. Similar to VAS-back, patients mark their level of pain on a horizontal line from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst imaginable pain". This scale is particularly important for evaluating radicular symptoms commonly associated with lumbar spinal stenosis.
Health-Related Quality of Life (EQ-5D-5L) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  The EQ-5D-5L questionnaire consists of two components: a descriptive system and a visual analog scale. The descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with five levels of problems each (no problems, slight problems, moderate problems, severe problems, extreme problems). The visual analog scale records the patient's self-rated health on a vertical scale where the endpoints are labeled 'the best health you can imagine' and 'the worst health you can imagine'. This tool has been validated for the Mexican population and allows derivation of the EQ-5D index value.
Patient Satisfaction with Surgical Outcomes (Modified MacNab Criteria) | 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure evaluates patient satisfaction with respect to functional outcomes obtained after undergoing the surgical procedure using the Modified MacNab Criteria. This scale has been widely used for decades as a tool to assess patient satisfaction and classifies outcomes as: Excellent (no pain or restriction of mobility, return to work and daily activities), Good (occasional non-radicular pain with symptom relief, able to return to work but with restrictions), Fair (some functional improvement, disability and/or inability to return to work), Poor (persists with radicular symptoms, requires new surgical intervention).
Duration of Hospitalization | Measured during the index hospitalization.
  This metric records the total number of days from patient admission until discharge following the surgical procedure. It serves as an indicator of the immediate postoperative recovery and overall efficiency of the surgical intervention.
Duration of Surgery | Recorded intraoperatively.
  This outcome measures the surgical time, defined as the period from the initial incision to the final closure of the surgical site. It reflects procedural efficiency and may indirectly indicate the technical ease or complexity of the procedure.
Intraoperative Blood Loss | Assessed during the surgical procedure.
  This measure quantifies the volume of blood lost during the surgical procedure, as collected via standard suction devices and measured in milliliters. It is an important indicator of surgical safety and efficiency.
Rate of Perioperative Complications | Assessed 7 days, 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure records the incidence and severity of complications occurring during the perioperative period. Complications will be categorized according to the Clavien-Dindo classification and summarized using the Comprehensive Complication Index, providing a quantitative assessment of overall surgical morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Benvenutti Regato, MD, Principal Investigator — TecSalud
Locations (1):
- Hospital Zambrano Hellion, TecSalud, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No